CLINICAL TRIAL: NCT00949078
Title: Effects of Omalizumab on Peanut Allergen Induced Cellular and Clinical Responses in Peanut Allergic Adults
Brief Title: Omalizumab in the Treatment of Peanut Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00026397; 1U19AI070345 (NIH)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Food Allergy; Peanut Allergy
Keywords: peanut; allergy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Label Omalizumab Group A (Experimental): Omalizumab was dosed according to package insert. Patients who have a decrease in peanut allergen induced basophil histamine release (Pn-BHR) to less than 20% of baseline will be assigned to this group.
  Interventions: Drug: omalizumab
- Open Label Omalizumab Group B (Experimental): Omalizumab was dosed according to package insert. Patients who do not have a decrease in peanut allergen induced basophil histamine release (Pn-BHR) to less than 20% of baseline will be assigned to this group.
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab — omalizumab subcutaneously every 2-4 weeks depending on participant weight and total IgE
  Other Names: Xolair

SUMMARY:
The purpose of this study is to determine if treatment with omalizumab (Xolair, anti-IgE) can eliminate or reduce symptoms of peanut allergy.

DETAILED DESCRIPTION:
The study will evaluate if omalizumab is an effective treatment for peanut allergy. In addition we will further evaluate the role of allergic cells (mast cells and basophils) and IgE in food allergy.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female (non-pregnant), age 18-50
* Females must be: Surgically sterile (hysterectomy, bilateral oophorectomy, bilateral tubal ligation), OR postmenopausal (at least 1 year since last menses), OR using one of the following medically acceptable forms of birth control throughout the duration of the study:

  * Systemic contraceptives
  * Diaphragm with intravaginal spermicide
  * Cervical cap
  * Intrauterine device
  * Condom with intravaginal spermicide Females in certain categories (not sexually active, vasectomized partner) will be admitted at the discretion of the investigator on a case-by-case basis.

Females, excluding those more than 1 year postmenopausal or who are surgically sterile, must have a negative urine pregnancy test at Visit 1 and other visits specified in this protocol. If a subject becomes pregnant during the study participation, they will be discharged from the study and followed for any adverse events until termination of the pregnancy or delivery is complete. Given that the drug is in pregnancy category B, we will follow the pregnant mother for any adverse events for the duration of the study.

* Physician diagnosed peanut allergy OR convincing clinical history of peanut allergy with its onset in early childhood.
* Positive puncture skin test to peanut greater than or equal to 3 mm diluent control
* Positive ImmunoCAP to peanut ≥0.35 kU/L.
* In vitro basophil responsiveness to peanut allergen, with greater than 20% histamine release or 10-19% if greater than 50% of an optimal anti-IgE response (at baseline visit).
* Subjects must have a positive oral food challenge to peanut as defined by having objective signs of a clear allergic reaction at a cumulative dose of peanut protein <1000 mg. Objective allergic signs may include oral urticaria, cutaneous urticaria, rhinorrhea, sneezing, coughing, wheezing, or vomiting.

Exclusion Criteria:

* Asthma with Forced Expiatory Volume in 1 second (FEV1) < 80% predicted or severe persistent asthma per National Asthma Education and Prevention Program (NAEPP) Standards (2007 National Asthma Education and Prevention Program Expert Panel Report III guidelines) or poorly controlled asthma with oral corticosteroid use for exacerbation in last 6 months.
* History of severe allergic reaction to peanut requiring intubation or ICU admission.
* Late onset peanut allergy, defined as subjects who had previously tolerated peanut on a regular basis before their initial reaction.
* Patients with biopsy proven eosinophilic enteropathy will be excluded.
* Patients with total serum IgE levels less than 30 IU/mL or greater than 700 IU/mL at the time of enrollment will be excluded.
* Patients with hematocrit < 32%, White Blood Cell (WBC) count <4000/microliter, platelet < 75000/microliter, creatinine > 141.4 micromolar/L, or Aspartate Aminotransferase (AST) > 100 IU/L will be excluded if these abnormalities are present at the time of enrollment.
* Body weight less than 30 kg or greater than 150 kg at enrollment will be excluded.
* Patients with plans to become pregnant or breastfeed will be excluded from the study. Patients must indicate they will use methods to avoid pregnancy.
* Other significant medical conditions (e.g., liver, gastrointestinal, kidney, cardiovascular, pulmonary disease, or blood disorders), which, in the opinion of the Investigator, make the subject unsuitable for induction of food reactions.
* Current or prior use of omalizumab in the past 12 months.
* Use of non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) or immunomodulator (not including corticosteroids) or biologic therapy within the past year.
* Use of beta-blockers (oral or ocular), angiotensin-converting enzyme (ACE) inhibitors, or angiotensin-receptor blockers (ARB) within 72 hours prior to either of the qualification Oral Food Challenge (OFC).
* Use of antihistamines (within 3 days for short acting and 5 days for long acting) prior to the screening OFC.
* Use of antihistamines (within 3 days for short acting and 5 days for long acting) prior to the study OFC. These procedures should be rescheduled when off antihistamines for the required time.
* Inability to discontinue antihistamines for routine study tests.
* History of ischemic cardiovascular disease (i.e., previous Myocardial Infarction, angina etc) or uncontrolled hypertension.
* Significant upper respiratory tract infection (URI) within 7 days of any OFC; OFCs should be rescheduled within 7 days following resolution of URI.
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
* Use of any investigational drugs within 8 weeks of participation.
* Any contraindication to omalizumab including patients with a previous hypersensitivity to omalizumab.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Wood, MD, Principal Investigator — Johns Hopkins University; Sarbjit Saini, MD, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Leung DY, Sampson HA, Yunginger JW, Burks AW Jr, Schneider LC, Wortel CH, Davis FM, Hyun JD, Shanahan WR Jr; Avon Longitudinal Study of Parents and Children Study Team. Effect of anti-IgE therapy in patients with peanut allergy. N Engl J Med. 2003 Mar 13;348(11):986-93. doi: 10.1056/NEJMoa022613. Epub 2003 Mar 10. PMID 12637608

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 participants underwent screening history and laboratory evaluation. Of those, 14 underwent a screening food challenge and were randomized to subsequent arms.
Period: Overall Study
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Decrease in Pn-BHR Area Under the Curve (AUC) of > 80% Compared With Baseline Values Before Week 8
Description: Presence or absence of this change
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 5 | 9
Participants | 5 | 9

2. Primary Outcome: Percent Change in Peanut Specific Immunoglobulin E (IgE) From Baseline to After Pn-BHR Response
Description: percentage
Time Frame: change from baseline to up to 6 months
Measure: Median (Full Range); unit: percentage change Peanut specific IgE
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 5 | 9
percentage change Peanut specific IgE | 1.9 [0.5 to 3.3] | 32 [3.3 to 41]

3. Primary Outcome: Peanut Specific Immunoglobulin E (IgE) After Pn-BHR Response
Description: kU/L (range)
Time Frame: up to 6 months
Measure: Median (Full Range); unit: kU/L
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 5 | 9
kU/L | 2.1 [1.1 to 13] | 30.5 [8.3 to 184]

4. Primary Outcome: Total Immunoglobulin E (IgE) After Pn-BHR Response
Description: kU/L (range)
Time Frame: up to 6 months
Measure: Median (Full Range); unit: kU/L
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 5 | 9
kU/L | 201 [110 to 523] | 129 [36 to 527]

5. Primary Outcome: Dose of Peanut Protein Inducing Allergic Symptoms at Oral Food Challenge (OFC) 1
Description: mg
Time Frame: up to 8 weeks
Measure: Median (Full Range); unit: mg
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 5 | 8
mg | 80 [30 to 380] | 80 [10 to 700]

6. Primary Outcome: Dose of Peanut Protein Inducing Allergic Symptoms at OFC 2
Description: mg
Time Frame: up to 8 weeks
Measure: Median (Full Range); unit: mg
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 4 | 9
mg | 6500 [3080 to 10000] | 6790 [180 to 100000]

7. Primary Outcome: Dose of Peanut Protein Inducing Allergic Symptoms at OFC 3
Description: mg
Time Frame: up to 8 weeks
Measure: Median (Full Range); unit: mg
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 4 | 6
mg | 8540 [1830 to 10000] | 2455 [1830 to 10000]

8. Primary Outcome: Omalizumab Received Before OFC 2
Description: Number of doses
Time Frame: up to 6 months
Measure: Median (Full Range); unit: number of doses
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 5 | 9
number of doses | 1 [1 to 3] | 3 [2 to 5]

9. Primary Outcome: Omalizumab Received Before OFC 2
Description: total mg
Time Frame: up to 6 months
Measure: Median (Full Range); unit: mg
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
Number analyzed (Participants) | 5 | 9
mg | 300 [300 to 675] | 900 [300 to 1875]

ADVERSE EVENTS:
Arm/Group | Open Label Omalizumab Group A | Open Label Omalizumab Group B
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes